CLINICAL TRIAL: NCT05183074
Title: Phase II Prospective Trial of MR-linac Based Stereotactic Ablative Radiotherapy for Patients With Localized (SAMRT-P01) and Oligo-metastatic (SMART-P02) Prostate Cancer
Brief Title: MR-linac Guided Ultra-hypofractionated RT for Prostate Cancer (SMART-P01 and SMART-P02)
Acronym: SMART-P01/02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NINGNING LU, Principle Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2277
Record Dates: First submitted 2021-12-02; First posted 2022-01-10 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Radiotherapy Side Effect; Magnetic Resonance-linac; Stereotactic Ablative RT; Adaptive Radiotherapy; Localised Disease; Oligometastatic Disease
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-linac group (Experimental): Pts received ultra-hypofractionated RT for primary w/o adjacent oligo-metastatic diseases on 1.5-Tesla MR-Linac
  Interventions: Device: MR-linac

INTERVENTIONS:
Device: MR-linac — 1.5-Tesla MR-linac based SBRT

SUMMARY:
1. To investigate the tolerability of MR-linac based stereotactic ablative radiotherapy (MRL-SBRT)for patients with localized prostate cancer
2. To assess the acute and late toxicities, efficacy and quality of life for patients treated by MRL-SBRT
3. To simulate the dose planning and assess the feasibility of simultaneous-boost for MR-prominent foci
4. To investigate the relationship between the changes of blood and tissue biomarkers and manifestations on mp-MRI pre-/post-MRL-SBRT, to further ascertain the predictive factors of local persisting and/or relapse disease

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years。
* Histology confirmed prostate cancer.
* Risk stratification, localised disease including patients with low-risk(cT1-T2a，PSA <10ng/mL，Gleason score≤6) who refuse active surveillance, favorable or unfavorable intermediate-risk and selected high-risk(cT2b-T3a or minimally T3b，PSA 10-40ng/mL，Gleason score 7-8) disease.
* Oligo-metastatic disease including patients with prostate in-situ and oligometastatic disease (no limit to mets number and organs, with all metastatic foci can be safely treated by radical SBRT dose)
* ECOG 0-2
* Postate gland volume ≤100cc
* IPSS score of <18
* Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed

Exclusion Criteria:

* Contraindications to MRI.
* TURP within the past 6 months
* Ulcerative colitis, Crohn's Disease, ataxia telangiectasia, or systemic lupus erythematosus
* Previous pelvic irradiation
* Refuse contraception

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Acute GU and GI toxicities: Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Three months post-MRL-SBRT
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
The Incidence of Late toxicities: Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 6-months, 1-year and 2-year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Quality of life evaluation | Every 2 weeks during SBRT and till 8 weeks after RT completion, every 3 months to 2 years and every 6 months to 5 years, and yearly thereafter
  Evaluate quality of life of patients by QOL questionnaires at different time points
Biochemical-relapse free survival | 2-year

CONTACTS AND LOCATIONS:
Locations (1):
- Radiotherapy Department of Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China